CLINICAL TRIAL: NCT04979117
Title: Diagnostic Performance of Superb Microvascular Imaging Ultrasonography in Plantar Fasciitis
Brief Title: Superb Microvascular Imaging Ultrasonography of Plantar Fasciitis
Acronym: SMI
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Ender Salbaş, Physical Medicine & Rehabilitation Specialist, MD, Nigde Omer Halisdemir University
Other Study IDs: ES01
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Diagnose Disease; Plantar Fasciitis
Keywords: superb microvascular imaging; diagnose; microvascularization; plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with plantar fasciitis: Participants with the diagnose of plantar fasciitis; typical anamnesis (exacerbating pain by the first steps in the morning or after rest and with prolonged standing).
  The emerge of local point tenderness over the heel and proximal fascia due to the pressure applied by the physician.
  Thickening of the plantar fascia greater than 4 mm in ultrasonographic evaluation. measurement
  Interventions: Device: Superb Microvascular Imaging (SMI) (Toshiba)
- Volunteers who has not foot complaints.: Volunteers who were not diagnosed with Plantar Fasciitis and without foot or heel pain when taking the first steps in the morning, with plantar fascia thickness less than 4 mm, painless, symptom-free and which had no additional rheumatic disease.
  Interventions: Device: Superb Microvascular Imaging (SMI) (Toshiba)

INTERVENTIONS:
Device: Superb Microvascular Imaging (SMI) (Toshiba) — to determine whether there is a diagnostic value of SMI in Plantar Fasciitis and whether there is a superiority when compared Power Doppler and Color Doppler modalities.

SUMMARY:
A prospective study will be conducted to evaluate the diagnostic performance of SMI, gray scale US, color Doppler US and Power Doppler US.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is a painful condition of the inferior and medial heel. Symptoms worsens with the first steps in the morning or after prolonged sitting and long periods of standing.

The diagnosis of PF is made according to the typical anamnesis and physical examination, based on the emerge of local point tenderness over the heel and proximal fascia due to the pressure applied by the physician. Heel pain exacerbates by the first steps in the morning or after rest and with prolonged standing. Unless there is an inflammatory disease such as spondyloarthropathy, there is no laboratory finding indicating plantar fasciitis. Imaging methods are very useful for making an accurate diagnosis. Because the main problem is in the soft tissue, plain radiography has limited diagnostic value, but can be helpful in identifying calcaneal stress fractures.

Magnetic resonance imaging (MRI) is very successful in showing the inflammatory process of soft tissue. However, it does not seem possible to use MRI scans routinely because of the cost and time it requires.

PF can be evaluated with ultrasonography with the advantages of being non-invasive, relatively inexpensive, easy to access and apply, and is increasingly used in clinical practice. Color Doppler evaluation is a very valuable part of musculoskeletal sonographic examination and facilitates the clinician's decision as an inflammation marker. Power Doppler US is quite sensitive to tissue or probe movement, especially at low pulsed repetition frequency (PRF). Flash artifacts may be observed. However, Doppler USG has limited sensitivity at low flows and small vessel structures.

Superb microvascular imaging (SMI) (Toshiba Medical Systems, Tokyo, Japan) is a new mode of vascular imaging that provides visualization of activity in microvascular structures or in structures that have low flow rate.

To the best of our knowledge, there are no studies comparing the diagnostic performance of the SMI modality in plantar fasciitis with color Doppler and gray scale US. Therefore, a prospective study will be conducted to evaluate the diagnostic performance of SMI, gray scale US, color Doppler US and Power Doppler US. The null hypothesis that there is no difference between Doppler US and SMI methods in the detection of increased inflammatory activity in plantar fasciitis patients.

ELIGIBILITY:
For the first group:

Inclusion Criteria:

* Patients who diagnosed as Plantar Fasciitis
* Age between 18-45

Exclusion Criteria:

* History of foot trauma or surgery
* Diabetes mellitus
* Pregnancy,
* Rheumatological diseases

For the second group:

Inclusion Criteria:

* asymptomatic foot,
* no previous trauma or surgery on foot,
* no history of systemic inflammatory disorders.

Exclusion Criteria:

* History of foot trauma or surgery
* Diabetes mellitus
* Pregnancy,
* Rheumatological diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Patients who diagnosed as Plantar Fasciitis as the first group
  * Healthy participants as the second group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | Each participant will be assessed only one time at the admission time to the outpatient clinic
  The patient will be asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line. This rating is then measured from the left edge gives the VAS score. A higher score indicates greater pain intensity and lower scores indicates less pain intensity.
Heel Tenderness Index (HTI) | Each participant will be assessed only one time at the admission time to the outpatient clinic
  Heel tenderness index (HTI) will be assessed by physician; based on assessing pain on palpation (0=no pain, 1=painful, 2=painful and winces, 3=painful, winces and withdraws).
Foot Function Index (FFI) | Each participant will be assessed only one time at the admission time to the outpatient clinic
  This index aims to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales.
Ultrasonographic Evaluation; Superb Microvascular Imaging, GrayScale Imaging, Color Doppler Imaging, Power Doppler Imaging | Each participant will be assessed only one time at the admission time to the outpatient clinic
  Vascular blood flow images from median nerve (enterrapted in carpal tunnel) obtained with Power Doppler and Superb microvascular imaging. [ Time Frame: Each participant will be assessed only one time at the admission time to the outpatient clinic ] Four-stage classify will be use for grading these images; Grade 0: No vascularity in MN, Grade 1: One or two focal color-encoded spots in MN, Grade 2: One linear color-encoded line or more than two focal color-encoded spots in MN, Grade 3: More than one linear color-encoded line in MN

CONTACTS AND LOCATIONS:
Overall Officials: Ender Salbas, MD, Study Director — Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not want to share IPD with any researchers.